CLINICAL TRIAL: NCT06720701
Title: Development of Prognostic Models for Response and Toxicity to CAR-T Cell Therapy in Patients with Relapsed/refractory Non Hodgkin's Lymphoma.
Acronym: CLIO
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CLIO; RC-2024-2790609 (Other Grant/Funding Number: Ricerca Corrente (Ministero della salute))
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Car-T therapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Observational, single-center, tissue-based cohort study involving both retrospective and prospective enrollment of patients undergoing CAR-T cell therapy and up to 1 year of prospective follow-up necessary to detect the outcomes required by the study

DETAILED DESCRIPTION:
This is a pharmacological observational study, with collection of biological material, single-centre, no-profit, involving both retrospective and prospective enrolment of patients undergoing CAR-T cell therapy and up to 1 year of prospective follow-up necessary to detect the outcomes required by the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with relapsed/refractory non-Hodgkin lymphoma, candidates to receive CAR-T cell therapy according to clinical indication
* Acquisition of informed consent for participation in the study
* Acquisition of consent to the processing of personal data.

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 125 patients who will participate in the study have been or are candidates to receive CAR-T cell therapy. CAR T therapy is intended as a therapeutic pathway.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Develop predictive models of response to CAR-T cell therapy at different time points in patients with relapsed/refractory non-Hodgkin lymphoma.. | 1,3 ,6 12 months post CAR-T therapy
  The outcome of objective 1 is the occurrence of one of the following conditions: complete response (CR) or partial response (PR) or stable response (SD) or progression of disease (PD). The outcome will be assessed by performing a PET/CT radiological examination.
  The response to treatment [(Overall Response Rate (ORR), or CR + PR] is defined as negativization of the uptake or Deauville score ≤3.
  The non-response to treatment/refractoriness [SD + PD] is defined as persistence/increase of the uptake, or Deuville Score >3.
Develop a predictive model of CRS toxicity to CAR-T cell therapy in patients with relapsed/refractory non-Hodgkin lymphoma | 7 days post CAR-T therapy
  The outcome of this objective is the occurrence of CRS toxicity events. The outcome will be assessed according to CTCAE vers. 5.0 CRS toxicity on treatment is defined as the incidence of CRS events of grade ≥1 and/or the incidence of ICANS of grade ≥1
Develop a predictive model of ICANS toxicity to CAR-T cell therapy in patients with relapsed/refractory non-Hodgkin lymphoma | +7 days post CAR-T infusion
  The outcome of this objective is the occurrence of ICANS toxicity events. The outcome will be assessed according to CTCAE vers. 5.0 ICANS toxicity on treatment is defined as the incidence of ICANS events of grade ≥1.

SECONDARY OUTCOMES:
To estimate the overall survival (OS) of patients with relapsed/refractory non-Hodgkin lymphoma who have undertaken the therapeutic pathway (i.e. from apheresis, by intention-to-treat) | 12 months post CAR-T infusion
  Death from any cause
To estimate the progression-free survival (PFS) of patients with relapsed/refractory non-Hodgkin lymphoma who have undertaken the therapeutic pathway (i.e. from apheresis, by intention-to-treat) | 12 months post CAR-T infusion
  disease status by PET/CT examination and defined as negative uptake or Deauville score ≤3.
To describe the characteristics of all therapy-related toxicity events (other than CRS and ICANS) in patients with relapsed/refractory non-Hodgkin lymphoma who received CAR-T cell therapy up to 12 months post-infusion. | untill 12 months
  Type, grade (according to CTCAE 5.0), onset date, end date, outcome

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No